CLINICAL TRIAL: NCT01440205
Title: Licensing Flu Shot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Katherine Milkman, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 813606-2
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Flu
Keywords: Flu Shot
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Easy list of healthy habits (Experimental): In this condition, participants will be prompted to think about a list of healthy behaviors and check off (privately - they will never send this flyer back or show it to anyone) whether "yes" they conform to the healthy habit or "no" they do not. The list of healthy behaviors is a list that most people will find fairly easy, and thus most participants will answer "yes" to each habit. The final question will be a prompt to get a flu shot. The hope is that when people realize how healthy their habits are, it will seem natural to them to engage in yet another healthy habit and receive a flu shot.
  Interventions: Behavioral: Easy list of healthy habits
- Challenging list of healthy habits (Experimental): In this condition, participants will be prompted to think about a list of healthy behaviors and check off (privately - they will never send this flyer back or show it to anyone) whether "yes" they conform to the healthy habit or "no" they do not. The list of healthy behaviors is a list that most people will find fairly difficult, and thus most participants will answer "no" to each habit. The final question will be a prompt to get a flu shot. The hope is that when people realize how unhealthy their habits are, it will seem wise to engage in one healthy habit that is easy (to make up for other bad behaviors) and receive a flu shot.
  Interventions: Behavioral: Challenging list of healthy habits
- Control (Experimental): A control condition with no list of healthy behaviors.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Easy list of healthy habits — The recipient will be prompted to check off "yes" or "no" to healthy habits that most people will find fairly easy.
  Arms: Easy list of healthy habits
Behavioral: Challenging list of healthy habits — The recipient will be prompted to check off "yes" or "no" to healthy habits that most people will find fairly difficult.
  Arms: Challenging list of healthy habits
Behavioral: Control — No check box element
  Arms: Control

SUMMARY:
The mailer will encourage all employees of one of Evive's partner companies to attend an on-site free flu shot clinic they are offering in the fall of 2011. The research will examine differences in follow-through on getting a flu shot at an on-site clinic among the targeted population during the ~1 month period when clinics are being offered (following the mailing) as a function of experimental condition.

ELIGIBILITY:
Inclusion Criteria:

* Employee at partner corporation

Exclusion Criteria:

* Employee already received a flu shot this season

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6098 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants that receive a flu shot | up to two months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States